CLINICAL TRIAL: NCT02154659
Title: The Difference of Reflux Pattern Between the Patients Who Have Postprandial Reflux Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2013-0680
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- postprandial reflux group (Other): Esophageal pH monitoring is the current gold standard for diagnosis of gastroesophageal reflux disease. It provides direct physiologic measurement of acid in the esophagus and is the most objective method to document reflux disease, assess the severity of the disease and monitor the reflux acidity.
  Interventions: Device: 24hr pH monitoring
- normal group (Other): Esophageal pH monitoring is the current gold standard for diagnosis of gastroesophageal reflux disease. It provides direct physiologic measurement of acid in the esophagus and is the most objective method to document reflux disease, assess the severity of the disease and monitor the reflux acidity.
  Interventions: Device: 24hr pH monitoring

INTERVENTIONS:
Device: 24hr pH monitoring

SUMMARY:
Gastroesophageal reflux disease is increasing worldwide. The causes of reflux symptoms are not found exactly. especially, the postprandial reflux symptoms are more common than the all day reflux symptoms. One of the causes of reflux symptoms is the relaxation of the lower sphincter of the esophagus. But, the sphincter relaxation also occur in normal people. But, there is a difference in postprandial reflux pattens between the patients and the normal people. So, in this study, we want to compare the difference of reflux pattern between the patients who have postprandial reflux symptoms and normal people though the 24hr pH monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. over 19 years old, male and female
2. normal people (control group, who has no postprandial reflux symptoms
3. patients who have postprandial reflux symptoms (postprandial reflux symptom means that within the last 6 months, postprandial reflux symptoms more than once a week for more than 1 month)

Exclusion Criteria:

1. patients who have nasoesophageal stricture
2. patients who have bleeding tendency
3. patients who have esophageal varix
4. patients who have cardioverter implantation
5. patients who had surgery for esophagus, stomach or duodenum
6. patients who are taking medications, gastrointestinal motility drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
The difference of reflux pattern at postprandial period between the patients who have postprandial reflux symptoms and the normal people | Within the 24 hours after the 24hr pH monitoring
  Primary Outcome - The difference of reflux pattern at postprandial period between the patients who have postprandial reflux symptoms and the normal people The postprandial reflux symptom means that the symptoms more than once for a week for more than 1 month

SECONDARY OUTCOMES:
The difference of esophageal reflux pH between the patients who have postprandial reflux symptoms and the normal people | Within the 24 hours after the 24hr pH monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university College of Medicine, Seoul, South Korea